CLINICAL TRIAL: NCT05202964
Title: Compliance and Tolerance to Oral AntiBiotherapy in Osteoarticular Infections
Brief Title: Compliance and Tolerance to Oral AntiBiotherapy in Osteoarticular Infections (OTABIO)
Acronym: OTABIO
Status: Recruiting | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL21_0905; 2021-A02134-37 (Other: ID RCB)
Record Dates: First submitted 2022-01-10; First posted 2022-01-24 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Drug-Related Side Effects and Adverse Reactions; Treatment Adherence and Compliance
Keywords: Tolerance; Adherence; Antibiotic; BJI; adverse effect
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions; Treatment Adherence and Compliance | interventions — Drug Tolerance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Tolerance and adherence to oral antibiotics in patients managed for BJI: Patients having a BJI treated by surgery and taking at least one oral antibiotic after the surgery
  Interventions: Other: Tolerance and adherence to oral antibiotics in patients managed for BJI

INTERVENTIONS:
Other: Tolerance and adherence to oral antibiotics in patients managed for BJI — Adherence will be measured 6 weeks (S6) and 3 months (M3) after the surgery. Tolerance will be mesured at baseline, and at 6 weeks (S6) and 3 months (M3) after the surgery.
  The compliance data collected will be compared by two methods (electronic pill dispensers and questionnaire).
  Patients will respond to a questionnaire about the tolerance of intraveinous antibiotics (between surgery and baseline) and oral antibiotics at baseline, and during the consultation at S6 and M3.
  Responses to the compliance questionnaire will be collected during a telephone interview by a member of the Croix-Rousse pharmacy at S6 and M3. The pill organizer data from S6 and M3 will be transferred to the software by a nurse.

SUMMARY:
Bone and joint infections (BJI) are most often bacterial infections that can occur after surgery or de novo. They are rarely fatal in the short term, but are associated with significant morbidity, impaired quality of life and significant costs. Treatment of BJI is based on antibiotic therapy, often combined with surgery. Antibiotic therapy, at high doses, lasts a minimum of 6 weeks. It can be responsible for severe adverse effects. These characteristics (prolonged duration, multiple daily doses, and adverse effects) are known to negatively affect treatment adherence in general.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years
* Diagnosis of osteoarticular infection
* Treatment with at least one oral antibiotic for a minimum expected duration ≥ 6 weeks with an expected end of treatment date
* Patient who was informed and did not object to participate in the study

Exclusion Criteria:

* Treatment for BJI with oral antibiotic without end of treatment date
* treatment for BJI with parenteral antibiotic only
* patient who doesn't have a telephone number or who doesn't want to give it
* Adults subject to a legal protection measure
* Pregnant or breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients having a BJI treated by at least one oral antibiotic after a surgery
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-06-13 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Percentage of doses taken at 6 weeks | At 6 weeks after surgery
  Ratio of the number of doses taken over the theoretical number of doses to be taken over the period
Percentage of doses taken at 3 months | at 3 months after surgery
  Ratio of the number of doses taken over the theoretical number of doses to be taken over the period

CONTACTS AND LOCATIONS:
Overall Officials: Valérie MIRABET, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Hospices Civils de Lyon, Lyon, France